CLINICAL TRIAL: NCT07054177
Title: Salivary Metabolomics of Pregnancy and Periodontal Disease Related Metabolic Pathways
Brief Title: Metabolic Profiling of Saliva in Pregnancy and Periodontal Disease
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E195935
Record Dates: First submitted 2025-06-25; First posted 2025-07-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Gingivitis and Periodontal Diseases
Keywords: pregnancy; gingivitis; periodontal disease; saliva; metabolomics; LC-MS/MS
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva samples will be collected from all participants during different stages of pregnancy (first, second, and third trimesters, and 6-8 weeks postpartum) and from non-pregnant healthy controls. The samples will be centrifuged and stored at -80°C until analysis. The retained specimens will be used solely for untargeted metabolomic analysis using LC-MS/MS. No DNA extraction or genetic testing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: This group includes 15 healthy pregnant women aged 18-40 with uncomplicated pregnancies. Saliva samples are collected at four time points: during the first (0-13 weeks), second (14-27 weeks), and third trimesters (28 weeks and later), and at 6-8 weeks postpartum. No medical intervention is applied. The aim is to analyze changes in periodontal parameters and salivary metabolite profiles over time using untargeted metabolomics via LC-MS/MS.
- Non-Pregnant Healthy Controls: This group includes 15 systemically healthy, non-pregnant women aged 18-40 with regular menstrual cycles and no history of pregnancy in the past 6 months. Saliva and periodontal measurements are collected during the early follicular phase of the menstrual cycle. These participants serve as the control group for comparative evaluation of salivary metabolomic profiles and periodontal health status.

SUMMARY:
This study aims to better understand how pregnancy affects the health of the gums and tissues that support the teeth. During pregnancy, hormone levels (like estrogen and progesterone) increase significantly. These hormonal changes can cause many changes in the body, including in the mouth. Some pregnant women may notice that their gums become swollen, red, or bleed more easily - this is called pregnancy gingivitis. It happens more often during the second and third trimesters and usually improves after birth. Even if a pregnant person has good oral hygiene, hormonal changes may still make the gums more sensitive to plaque and bacteria. Scientists believe that these changes in gum health are linked to how the body responds to hormones, bacteria in the mouth, and changes in the immune system. To explore this further, saliva samples will be collected from:

* Pregnant women during their 1st, 2nd, and 3rd trimesters
* The same women again 6-8 weeks after giving birth
* A group of non-pregnant, healthy women as a comparison group The investigators will use a scientific method called untargeted metabolomics to study these saliva samples. This method helps looking at small substances (called metabolites) in saliva to see if there are any patterns related to pregnancy and gum health.

The goal is to identify biological changes that happen during pregnancy and understand how they might affect the gums. This research will help improve early detection and prevention of gum problems during pregnancy in the future.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the impact of physiological hormonal changes during pregnancy on periodontal status and to determine the metabolic pathways through which this effect occurs. For this purpose, saliva samples collected at different stages of pregnancy (1st, 2nd, and 3rd trimesters), in the postpartum period, and from systemically healthy non-pregnant individuals will be analyzed using an untargeted metabolomic approach based on LC-MS/MS. The analysis aims to identify potential metabolites and biochemical pathways that reflect the relationship between pregnancy-associated hormonal changes and periodontal tissues, thereby contributing to a better understanding of the underlying biological mechanisms.

This study will include 15 volunteer pregnant women aged 18-40, who are systemically healthy and whose pregnancy is progressing without complications, followed by a single gynecologist at the Department of Obstetrics and Gynecology, Bezmialem Vakıf University. The diagnosis of pregnancy will be confirmed by the detection of positive serum beta-hCG (human chorionic gonadotropin) levels and ultrasound confirmation of intrauterine gestation. Trimesters will be clearly classified according to gestational week determined by ultrasound. The included participants will be followed in the 1st (weeks 0-13), 2nd (weeks 14-27), and 3rd trimesters (week 28 and later), as well as at 6-8 weeks postpartum.

The control group will consist of 15 systemically healthy volunteers aged 18-40, who apply to the Department of Periodontology at Bezmialem Vakıf University. These participants will have a regular menstrual cycle, no hormonal disorders or systemic diseases, and no pregnancy within the last six months. Informed consent will be obtained from all participants before enrollment. Medical and dental histories will be recorded at the beginning of the study.

To evaluate periodontal status, plaque index (PI), bleeding on probing (BOP), probing depth (PD in mm), and clinical attachment level (CAL) will be measured at each visit (1st, 2nd, and 3rd trimesters and postpartum period for pregnant women, and early follicular phase of spontaneous or progesterone-induced menstrual cycle for controls). All measurements will be performed by a single calibrated periodontist at the Department of Periodontology, Bezmialem Vakıf University. Periodontal parameters will be recorded at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual) using a Williams periodontal probe (Hu-Friedy, Chicago, IL). Third molars will be excluded.

Participants with no clinical attachment loss, probing depth ≤3 mm, and bleeding on probing <10% will be classified as periodontally healthy. Those with no clinical attachment loss, probing depth ≤3 mm, and BOP >30% will be considered as having gingivitis. Participants with interproximal clinical attachment loss on at least two non-adjacent teeth and probing depth ≥4 mm will be diagnosed with periodontitis. Oral hygiene instructions will include the use of mechanical aids only (toothbrush, dental floss, interdental brush), and participants will be instructed to avoid using mouthwash or antimicrobial agents.

Before clinical periodontal measurements, saliva samples will be collected by another periodontist. Participants will be instructed not to eat or drink anything (except water) and not to chew gum before sampling, following an overnight fast. Unstimulated saliva will be collected by asking the participant to pool saliva in the mouth for approximately 5 minutes and then gently spit approximately 2.0 mL of saliva into a sterile glass beaker. The samples will then be transferred to sterile Eppendorf tubes using a micropipette, labeled, and stored at -80°C until analysis.

Before analysis, all saliva samples will be centrifuged at +4°C, 10,000 g for 10 minutes by a single researcher at the Department of Medical Biochemistry, Bezmialem Vakıf University, to remove particulate matter. The samples will then be prepared for LC-MS/MS analysis. In the LC-MS/MS system, each sample will first be separated into components by liquid chromatography (LC) and then identified based on their molecular masses using mass spectrometry (MS).

The data obtained from mass spectrometry will be analyzed using metabolite identification software and international metabolite databases (HMDB, KEGG, METLIN, etc.). The resulting metabolomic profiles will be used to explore biological pathways associated with pregnancy and periodontal status.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* No history of systemic disease or chronic infection
* No use of antibiotics or anti-inflammatory drugs in the last 3 months
* Non-smoker and non-alcohol user
* Willingness to participate by signing the informed consent form

Additional Criteria for Pregnant Volunteers:

* Singleton pregnancy (no multiple gestation)
* Pregnancy progressing without complications (e.g., no diagnosis of preeclampsia, gestational diabetes, or threatened preterm labor)
* Gestational age confirmed by ultrasound

Additional Criteria for Non-Pregnant Control Group:

* No history of pregnancy in the past 6 months
* Regular menstrual cycles
* No history of hormonal disorders (e.g., polycystic ovary syndrome, thyroid dysfunction)

Exclusion Criteria:

* Use of anti-inflammatory or antimicrobial treatments in the past 3 months
* Smoking or alcohol consumption
* Body mass index (BMI) > 30 kg/m²
* Presence of systemic diseases including diabetes mellitus, hyperprolactinemia, congenital adrenal hyperplasia, androgen-secreting tumors, thyroid dysfunction, Cushing's syndrome, hypertension, liver or kidney dysfunction
* Use of medications that may affect metabolic or hormonal parameters, such as oral contraceptives, steroid hormones, antihypertensives, or insulin-sensitizing drugs
* Periodontal treatment in the past 6 months
* Use of medications known to affect periodontal status (e.g., phenytoin, calcium channel blockers, cyclosporine, warfarin, NSAIDs, aspirin > 81 mg)
* Active infectious diseases such as hepatitis, HIV, or tuberculosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals assigned female at birth are eligible to participate, as the study focuses on pregnancy and related hormonal and periodontal changes.
Study Population: The study population includes systemically healthy pregnant women in different trimesters and postpartum period, and non-pregnant healthy women aged 18-40 years attending routine gynecology or periodontology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Salivary Metabolite Profile by Pregnancy Status | Baseline, 1st trimester (0-13 weeks), 2nd trimester (14-27 weeks), 3rd trimester (28 weeks and later), and 6-8 weeks postpartum
  Untargeted metabolomic analysis of saliva samples will be performed using LC-MS/MS to identify metabolite patterns associated with different stages of pregnancy and periodontal status. Results will be reported as relative metabolite concentrations (normalized intensity, arbitrary units).

SECONDARY OUTCOMES:
Bleeding on Probing (BOP) | Baseline, 1st trimester (0-13 weeks), 2nd trimester (14-27 weeks), 3rd trimester (28 weeks and later), and 6-8 weeks postpartum
  Bleeding will be recorded at six sites per tooth using gentle probing. The outcome will be reported as the percentage of bleeding sites per participant.
Plaque Index score | Baseline, 1st trimester (0-13 weeks), 2nd trimester (14-27 weeks), 3rd trimester (28 weeks and later), and 6-8 weeks postpartum
  Plaque accumulation will be assessed using the Silness-Löe Plaque Index (range: 0-3). The mean plaque index score per participant will be reported.
Mean probing depth (PD) | Baseline, 1st trimester (0-13 weeks), 2nd trimester (14-27 weeks), 3rd trimester (28 weeks and later), and 6-8 weeks postpartum
  Probing depth will be measured in millimeters (mm) at six sites per tooth. The average probing depth per participant will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Faculty of Dentistry and Faculty of Medicine, Istanbul, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided